CLINICAL TRIAL: NCT05681897
Title: Comparing Platelet-Rich Plasma (PRP) Centrifugation Methods on Thrombocyte Concentration and Clinical Improvement of Androgenetic Alopecia: A Preliminary, Randomized, Double-Blind Clinical Trial
Brief Title: Comparing Platelet-Rich Plasma (PRP) Centrifugation Methods on Thrombocyte Concentration and Clinical Improvement of Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Lili Legiawati, SpKK(K), National-board certified dermatologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 876/UN2.F1/ETIK/PPM.00.02/2
Record Dates: First submitted 2022-12-20; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Alopecia, Androgenetic
Keywords: Androgenetic Alopecia; Centrifugation; Platelet-rich plasma; Thrombocyte
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: this is a double-blind masking study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Spin Group (Other): Currently, the standard operating procedures for PRP preparation in dr. Cipto Mangunkusumo National General Hospital is by performing a single-spin centrifugation at 3000 rpm for 15 minutes. This first group will received PRP treatment by single-spin centrifugation at 3000 rpm in 15 minutes in addition to topical minoxidil (5%)
  Interventions: Procedure: Platelet-Rich Plasma Injections (PRP) on the Scalp
- Double Spin Group (Active Comparator): This group will received double-spin centrifugation PRP treatment at 1500 rpm in 6 minutes and continued at 2500 rpm in 15 minutes in addition to topical minoxidil (5%)
  Interventions: Procedure: Platelet-Rich Plasma Injections (PRP) on the Scalp

INTERVENTIONS:
Procedure: Platelet-Rich Plasma Injections (PRP) on the Scalp — each subject will be treated with 3x PRP injections on the scalp with 2 weeks interval in addition to daily minoxidil administration.
  Other Names: Regrou Forte (5% Minoxidil solution)

SUMMARY:
This research is a preliminary, randomized, double blind clinical trial, which will examine the differences in PRP preparation methods, a single-spin centrifugation of 3000 rpm in 15 minutes compared to a double-spin centrifugation of 1500 rpm in 6 minutes followed by 2500 rpm in 15 minutes, on the results of Thrombocyte Concentration and Clinical Improvement of Androgenetic Alopecia.

DETAILED DESCRIPTION:
Several examinations will be performed in every visit, including history taking, physical examination, trichoscopy and trichoscan. Laboratory evaluations (complete blood count) for the measurement of the thrombocyte for baseline and PRP will be performed for all assented subjects on the first visit. Each subject will be instructed to apply 5% topical minoxidil twice a day everyday as primary therapy during the study

ELIGIBILITY:
Inclusion Criteria:

* Met the criteria of androgenic alopecia (Hamilton Norwood grade III-IV)
* Men between ages 25-59 years old
* Have stopped taking topical anti-androgen or minoxidil for at least one month, or oral anti-androgen or minoxidil for at least three months

Exclusion Criteria:

* alopecia of any other type
* subject with a history of keloid or blood coagulation disorders underwent anticoagulant therapy
* subjects on Non-Steroidal Anti-Inflammatory Drugs (NSAID) medications in seven days prior to the study
* subjects who had hair treatment using growth factors, including PRP and microneedling within at least six months prior to the study.

Ages: 25 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 30 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Thrombocyte Count in PRP and Whole Blood | 6 weeks
  We assessed the increase in PRP platelet levels by assessing baseline platelets (using whole blood) and assessing platelet levels in PRP preparations and then calculating multiples. platelet valuie units to be used is (/μL)
Clinical Improvement of Androgenetic Alopecia | 6 weeks
  We assessed the assessment of clinical improvement in androgenetic alopecia using trichoscopy and trichoscan examination on week 0, 2, 4, and 6. On trichoscopic examination we assessed hair color, hair diameter diversity, vellus hair, and dots. Whereas on trichoscan examination we assessed hair count, hair diameter (mm), hair density (/cm2), hair rate (%) in vellus hair, terminal, anagen and telogen phases and assessed hair mean thickness (mm/cm2) and mean length (mm) and average hair per unit.

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta
  - Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region

REFERENCES:
- [Derived] Legiawati L, Yusharyahya SN, Bernadette I, Novianto E, Priyanto MH, Gliselda KC, Iriyanty S, Mutiara R. Comparing Single-spin Versus Double-spin Platelet-rich Plasma (PRP) Centrifugation Methods on Thrombocyte Count and Clinical Improvement of Androgenetic Alopecia: A Preliminary, Randomized, Double-blind Clinical Trial. J Clin Aesthet Dermatol. 2023 Dec;16(12):39-44. PMID 38125672